CLINICAL TRIAL: NCT04746612
Title: A Phase I, Multi-centre, Open-Label, First in Human Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of HH30134 in Patients With Advanced Solid Tumours
Brief Title: First in Human Study to Evaluate the Safety, Tolerability of HH30134 in Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor business decision
Sponsor: Haihe Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HH30134-G101
Record Dates: First submitted 2021-01-19; First posted 2021-02-10 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2022-12

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HH30134 (Experimental): HH30134 administered orally on a continuous once daily(QD), start from 100mg QD.
  Interventions: Drug: HH30134

INTERVENTIONS:
Drug: HH30134 — HH30134 administered orally on a continuous once daily(QD) in patients with advanced solid tumors

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics (PK), and to determine the maximum tolerable dose (MTD) and/or recommended phase 2 dose (RP2D) of HH30134 administered orally on a continuous once daily (QD) schedule in adults patients with advanced solid tumors.

DETAILED DESCRIPTION:
Study population

This is a global study involving multi-countries and multi-sites. Approximately 60 patients will be enrolled from participation institutions from different countries.

Enrollment in dose-escalation phase must have histologically or cytologically confirmed advanced solid tumors that have recurred or progressed following the last line of therapy and at least one prior standard of care regimens, or tumor for which there is no approved therapy, or for which standard therapy is unsuitable or refused. Enrollment in dose-expansion phase will be patients with selected solid tumors including but not limited to NSCLC and mCRC.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form.
* Stated willingness to comply with all study procedures and availability for the duration of the study.
* Male and female patients ≥ 18 years of age (or having reached the age of majority according to local laws and regulations, if the age is > 18 years)
* Patients must have histologically or cytologically confirmed advanced solid tumors
* Predicted life expectancy of ≥ 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
* Availability of archival tissue within three years or fresh tumor biopsy sample
* Patients must have adequate hepatic and renal function

Exclusion Criteria:

* Patient has received any anticancer therapy (including chemotherapy, targeted therapy, hormonal therapy, biotherapy, immunotherapy, or other investigational agents.) within 28 days or 5 times of half-lives (whichever is shorter) prior to the first dose of the study treatment.
* Radical radiation therapy (including radiation therapy for over 25% bone marrow) within 4 weeks prior to the first dose of the investigational product or received local palliative radiation therapy for bone metastases within 2 weeks.
* Any toxicities from prior treatment that have not recovered to baseline or ≤ CTCAE v5.0 Grade 1 before the start of study treatment, with exception of hair loss.
* Patients who have symptomatic CNS metastasis which is neurologically unstable or those who have CNS disease requiring increase in the dose of steroid.
* Major surgery or had significant traumatic injury within 28 days prior to the first dose of the investigational product or has not recovered from major side effects.
* Known HIV infection with a history of acquired immunodeficiency syndrome (AIDS)- defining opportunity infection within the past 12months; active hepatitis B and hepatitis C. Patients whose test results meet one of the following will not be enrolled:
* Patient is currently receiving or has received systemic corticosteroids ≤ 2 weeks prior to starting study treatment, or who have not fully recovered from side effects of such treatment.
* Gastrointestinal condition which could impair absorption of study medication.
* Patients with clinically significant cardiovascular disease
* Any diseases or medical conditions, at the Investigator's discretion, that may be unstable or influence their safety or study compliance, including organ transplantation, abuse of psychotropic medication, alcohol abuse or history of drug abuse.
* Other serious illness or medical conditions at the Investigator's discretion, that may influence study results, including but not limited to serious infection, diabetes, cardiovascular and cerebrovascular diseases or lung disease.
* Pregnant or breast-feeding patients. Pregnancy refers to the state of a woman between fertilization and the end of pregnancy confirmed by a positive laboratory hCG test (> 5 mIU/mL). Breast-feeding woman can become eligible for this study if she stops breast-feeding, however, cannot restart the breast-feeding on/after the completion of the study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-04-08 (Actual); Primary Completion 2023-03-24 (Actual); Study Completion 2023-03-24 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicities(DLT) | 12 months
  Incidence rate of dose limiting toxicities(DLT)
Maximum Tolerated Dose | 12 months
  To determine the maximum tolerable dose

SECONDARY OUTCOMES:
Pharmacokinetic(PK) measures - Plasma concentration-time Area Under the Curve | 12 months
  Measure the HH30134 concentration in blood plasma as a function of time
Pharmacokinetic(PK) measures - Cmax | 12 months
  Measure the maximum plasma concentration of HH30134
Pharmacokinetic(PK) measures - Tmax | 12 months
  Measure of time to reach maximum plasma concentration after administration of HH30134
Pharmacokinetic(PK) measures - CL/F | 12 months
  Measure apparent total clearance of HH30134 from plasma after administration
Pharmacokinetic(PK) measures - Vz/F | 12 months
  Measure apparent volume of distribution during terminal phase after administration of HH30134
Pharmacokinetic(PK) measures - terminal half-life(T1/2) | 12 months
  Measure elimination half-life of HH30134

CONTACTS AND LOCATIONS:
Overall Officials: Yaling QI, Study Director — Haihe Biopharma
Locations (4):
- Australia (2):
  - Blacktown Hospital, Blacktown
  - Scientia Clinical Research, Randwick
- China (2):
  - Sun Yat-sen University Cancer Center, Guangzhou
  - Fudan University Zhongshan Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No